CLINICAL TRIAL: NCT03345173
Title: Glutamatergic Modulation to Facilitate Naltrexone Initiation: A Randomized, Controlled Trial
Brief Title: Facilitating Rapid Naltrexone Initiation
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elias Dakwar, Research Scientist, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7543; 5R01DA042070-04 (NIH)
Record Dates: First submitted 2017-11-13; First posted 2017-11-17 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CI-581a (Experimental): CI-581a will be administered during the washout phase when participants are experiencing moderate withdrawal, as well as the following day when the naltrexone titration is initiated.
  (0.11 mg/kg 2-min bolus followed by 1.3 mg/kg over 90 min)
  Interventions: Drug: CI-581-a
- CI-581b (Placebo Comparator): CI-581b will be administered during the washout phase when participants are experiencing moderate withdrawal, as well as the following day when the naltrexone titration is initiated.
  (2-min saline bolus followed by 0.0125 mg/kg over 90 min)
  Interventions: Drug: CI-581-b

INTERVENTIONS:
Drug: CI-581-a — Two infusions in the context of naltrexone induction protocol.
  Arms: CI-581a
Drug: CI-581-b — Two infusions in the context of naltrexone induction protocol.
  Arms: CI-581b

SUMMARY:
The incidence of opioid use disorders (OUDs) has increased to near-epidemic proportions. While maintenance with long-acting opioids such as methadone or buprenorphine represents an effective treatment strategy, it may be unacceptable to many individuals. As a result, long-acting injectable naltrexone (XR-NTX), an antagonist medication that blocks the effects of opioids for at least 4 weeks, is now indicated for relapse prevention following detoxification. This randomized, controlled trial aims to test the efficacy of a glutamate modulator at facilitating a rapid non-opioid based naltrexone induction.

DETAILED DESCRIPTION:
This study combines a nonopioid detoxification; a naltrexone titration schedule that allows for pushing the dose rapidly while monitoring closely to ensure tolerability; and infusions integrated into the treatment in such a way as to potentially ameliorate spontaneous and precipitated withdrawal. The first part of the treatment trial involves receiving inpatient treatment for up to 5 days. Following week 1, participants will meet with staff twice weekly and receive 12 weeks of mindfulness based relapse prevention and motivational interviewing sessions.

ELIGIBILITY:
Inclusion Criteria:

1. DSM-5 criteria of current opioid use disorder present for at least six months, supported by a positive urine for opioids or a positive naloxone challenge test
2. Aged 18 to 70 years
3. In otherwise good health based on complete medical history, physical examination, vital signs measurement, ECG, and laboratory tests (hematology, blood chemistry, urinalysis) within normal ranges
4. Able to give written informed consent to participate in the study
5. Interested in maintenance treatment with extended-release naltrexone

Exclusion Criteria:

1. Physiologically dependent on alcohol or sedative-hypnotics with impending withdrawal requiring medical management
2. Methadone maintenance treatment or regular use of illicit methadone (>30 mg per week); urine toxicology positive for methadone at admission
3. Buprenorphine maintenance treatment or regular use of buprenorphine (>16 mg per week); urine toxicology positive for buprenorphine at admission
4. Active, or past, psychiatric disorder(s) which might interfere with participation or make participation hazardous, including DSM-V mental disorder due to another medical condition, major depressive disorder, psychotic disorder, or bipolar disorder with psychotic features
5. Significant current suicidal risk or a suicide attempt within the past year
6. On psychotropic or other medications that may interact adversely with study medications, or whose effect might be disrupted by study medications
7. For women of childbearing potential: positive serum pregnancy test, lactation, or unwillingness to use a satisfactory method of birth control
8. Unstable physical disorders which might make participation hazardous such as hypertension (>160/90), anemia, active hepatitis or other liver disease (transaminase levels < 2-3 X the upper limit of normal will be considered acceptable), or untreated diabetes. Participants reporting HIV+ status will be asked to provide information about their current treatment, including all medications. Participants who are on the antiretroviral ritonavir (Norvir) will be excluded due to the possibility that the study medications in combination with this medication may increase the risk of drug-induced hepatitis
9. Acute hepatitis with SGOT or SGPT > 3 times the upper end of the laboratory normal range
10. Concurrent participation in another treatment study or another substance abuse program with the exception of a self-help group
11. History of allergy or sensitivity to any study medication
12. Ongoing chronic pain that may require opioid management, or for which surgery is indicated
13. History of inability to tolerate study medications
14. History of a use disorder with the study medications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-11-25 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
XR-NTX Initiation | From baseline to week 12
  Initiation of XR-NTX during the inpatient induction, without dropout or buprenorphine initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Elias Dakwar, MD, Principal Investigator — NYSPI
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States